CLINICAL TRIAL: NCT02952456
Title: Phenomenological Approach of Epilepsy in Patients With Epilepsy and Their Relatives for Risk Prevention
Brief Title: Phenomenological Approach of Epilepsy in Patients With Epilepsy
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Université Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: UF9682
Record Dates: First submitted 2016-10-31; First posted 2016-11-02 (Estimated); Last update posted 2022-08-11 (Actual); Status verified 2022-08

CONDITIONS: Epilepsy
Keywords: SUDEP; Epilepsy; Qualitative research; Risks associated with epilepsy; Epilepsy-related deaths
MeSH Terms: conditions — Epilepsy; Sudden Unexpected Death in Epilepsy | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Bereaved families: Person who have lost a loved one from an epilepsy-related death with interview with a psychologist
  Interventions: Other: interview with a psychologist
- Patients with épilepsy: Patients with épilepsy with interview with a psychologist
  Interventions: Other: interview with a psychologist
- Relatives of patients with epilepsy: Relatives (Parents / spouse/ Husband) of patients with epilepsy with interview with a psychologist
  Interventions: Other: interview with a psychologist

INTERVENTIONS:
Other: interview with a psychologist — interview with a psychologist in Bereaved families, Patients with épilepsy and relatives of patients with epilepsy Relatives (Parents / spouse/ Husband) of patients with epilepsy

SUMMARY:
Rationale : Persons with epilepsy have a greater risk of incurring accidental injury and a higher mortality risk than the general population.

The main objective of the study is to understand life experience of the disease or risks associated with epilepsy in patients with epilepsy, relatives of patients and bereaved families.

Study design: Qualitative study (study based on interviews) Population: Three groups will be interviewed: bereaved families, patients with epilepsy and relatives of patient. Bereaved family: relatives who contact the French sentinel network "Réseau Sentinelle Mortalité Epilepsie" (RSME) notifying an epilepsy-related death (regardless the cause of the death and the timeframe between death and interview). Patients with epilepsy: patients having a secure diagnostic of epilepsy from 15 years old to 65 years old. Relatives of patients with epilepsy: spouse/husband or parents invited by a patient with epilepsy to participate to the interview who consent to participate.

Method: Semi structured in-depth interviews will be conducted by an experienced qualitative psychologist in face to face, at home, at the hospital or at any other place (depending on the choice of the participants). The interview topic guide will be centered on participants'personal experience. Interviews will be digitally recorded and will be transcribed by a secretary.

The results of this study will be integrated in educational therapeutic programs regarding prevention of risks related to epilepsy.

DETAILED DESCRIPTION:
Rationale: Persons with epilepsy have a greater risk of incurring accidental injury and a higher mortality risk than the general population.

Study Objective : To understand life experience of the disease and risks associated with epilepsy in patients with epilepsy, relatives of patients with epilepsy and bereaved families.The results of this study will be integrated in educational therapeutic programs regarding risks related to epilepsy.

Study design : Qualitative study with a phenomenological approach and semiopragmatic analysis. Three different groups will be interviewed: bereaved families, patients with epilepsy and relatives of patients with epilepsy.

Recrutement procedures :

The identification of bereaved families will be based on the French sentinel network "Réseau Sentinelle Mortalité Epilepsie" (RSME). This network was initially established by the French League Against Epilepsy (LFCE) under the leadership of bereaved families in 2010 and supported by the French Foundation for Epilepsy Research (FFRE). The primary aim of the RSME is to detail the causes and circumstances of epilepsy-related deaths in France. Secondary objectives are to evaluate the expectations and needs of bereaved families and create a national database for future research programs. Epilepsy-related deaths are reported by physicians but also by bereaved families. The interview will be proposed at this moment. Moreover the RSME includes a national network of bereaved families. The interview will be also proposed to the participants of this network.

Patients with epilepsy will be recruited from tertiary epilepsy units, private neurologists or general practitioners and thanks from patients associations. Patients living in the Languedoc Roussillon area and referred to the epilepsy unit of the University Hospital of Montpellier (CHRU Montpellier) will be preferentially invited to participate to the interview. The interview will be also proposed to relatives of patients (parents or spouse/husband) who consent to participate. The study could be proposed to patients included in the PRERIES study (Risk Factors in Sudden Unexpected Death in Epilepsy: A matched case-control study, coordinated by the coordination unit of the RSME).

Method :The characteristics of this methodology are based on COREQ criteria (consolidated criteria for reporting qualitative research).

A qualitative study with phenomenological approach will be used. The aim of this approach is to collect participants 'life-experiences in their own real and personal situation. Semistructured interviews with an in-depth questioning will be conducted by a psychologist who received specific patient-centered interview training. The interview topic guide using open questions will be centered on participants' personal experience.The same topic guide will be used for the first group (epileptic patients) and the second group (relatives group). However, for the third group (bereaved families), the interview guide will be adapted, looking at life experience before death: focusing circumstances, particular events, behaviors or clinical signs which could give alarm. This interview is more difficult because of a frequent sense of guilt and requires an experienced qualitative interviewer.The phenomenological questions will be asked on a temporal prospect.The first part, concern the disclosure of the disease. The questions invite participants to relive this moment, remembering when they were told about epilepsy and what happened after that: how they felt, what they thought? Behaviors and how the risks of epilepsy were be told by doctors.Secondly, participants will be invited to describe the current disease influence on the way of life.The key topics guide focused on epilepsy influence on body, relation to others or to relatives, employment, lifestyle and personal identity.

The saturation point will be determined when no more new information pertaining to the matter of research emerge.

The interviews will be conducted in face to face at home, at the hospital or in any other place (depending on the choice of the participants). The different conditions in which the interviews will be conducted will be all clearly identified and included in each recording: time, place, positioning of the actors, and context (family presence, disturbing environment). Interviews will be digitally recorded and will be transcribed by a secretary. According to that comprehensive approach, categories will be not identified in advance but derived from the data.

Other data collected : Sociodemographic data (gender, age, current occupation, education level, leasure, physical activity, driving and lifestyle) will be collected from a questionnaire filled in by the participants before the interviews. Clinical characteristics (duration of epilepsy, age at onset, syndrome and etiology, seizure type, seizures frequency) will be completed by the physicians in charge of the patients. For bereaved families, the cause of death will be recorded.

Data analysis :

Sample size : In qualitative studies, the sample size cannot be determined previously. Patients or relatives who satisfy the inclusion criteria will be invited for the study participation until a saturation point.

The saturation point is determined as the point at which further collection of data does not result in uncovering any new information pertaining to the topic under investigation. We estimate that approximately 30 interviews would be sufficient to reach data saturation.

Transcripts analysis : The analysis will be conducted using a grounded theory approach incorporating the pragmatism of Peirce. A semiopragmatic analysis according to CS Peirce's theories (semiopragmatical approach) guarantees a clearly and precise analysis and limits the biases or errors of interpretation. So, conceptual categories will not be identified not in advance but will be derived from the data by constant comparison.

Transcripts will be analyzed by two qualitative methodologists following these steps:Transcribing the recordings word for word (verbatim), Floating reading then focused reading, Breaking the text down into units of meaning and themes, Identifing all the semiotic, textual and contextual elements to let the category emerge through constant comparison (empirical category), Characterizing the empirical categories obtained according to the theory of classes of Signs (semiotics) (Quality, Fact, Law), Setting the categories in hierarchical order according to relationships between them in which law presuppose fact who presuppose quality, econstructing the meaning in the form of a synthetic generalizing proposition to restore the meaning of studied phenomenon Verbatim extract will be presented to illustrate the obtained categories with a number in order to identify them anonymously.

Descriptive analysis: Descriptive statistics on sociodemographic and clinical characteristics will be performed using SAS® version 9.1. (SAS Institute, Cary, NC). Intergroup differences will be examined using chi-squared and Mann-Whitney U analyses.

Practical course Study procedures and visits Informed consent procedures :The participant or participant's parent(s) / legal representative(s) must be informed by the interviewer about all aspects of the study that are relevant to decide to participate in particular concerning the personal data collection, and must have sufficient time and opportunity to ask any questions. Prior to the interviews, the written Informed Consent form must be signed and personally dated by the participant or participant's parent(s) / legal representative(s).

Collection of data: This interview will be conducted by a psychologist using the interview topic guide and a standardized form for sociodemographic data and clinical data.

ELIGIBILITY:
Inclusion Criteria:

* Bereaved family: Parents or spouse/husband who contact the coordination unit of the RSME in order to notify an epilepsy related death and who consent for an interview regardless of the cause of death and timeframe between death and interview.
* Patients with epilepsy: Patients having a secure diagnostic of epilepsy with active epilepsy (treated or not) or in remission under treatment or without treatment aged from 15 years to 65 years old.
* Relatives of patients with epilepsy: Parents or spouse/husband invited by a patient with epilepsy to participate to the interview who consent to participate.

Exclusion Criteria:

* Patients or relatives with learning difficulties
* Refusal of participation of the patients or relatives or legal representatives for patients aged under 18 years old
* Refusal for audio recording

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The identification of bereaved families will be based on the French sentinel network "Réseau Sentinelle Mortalité Epilepsie". This network was initially established by the French League Against Epilepsy under the leadership of bereaved families in 2010 and supported by the French Foundation for Epilepsy Research . The primary aim of the RSME is to detail the causes and circumstances of epilepsy-related deaths in France. Secondary objectives are to evaluate the expectations and needs of bereaved families. Epilepsy-related deaths are reported by physicians but also by bereaved families. The interview will be proposed at this moment. Moreover the RSME includes a national network of bereaved families. The interview will be also proposed to the participants of this network.Patients with epilepsy and relatives of patients will be recruited from tertiary epilepsy units, private neurologists or general practitioners and thanks from patients associations.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2016-09; Primary Completion 2017-11 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
interview with a psychologist | 1 day
  The aim of this approach is to collect participants 'life-experiences in their own real and personal situation. Semistructured interviews with an in-depth questioning will be conducted by a psychologist The interview topic guide using open questions will be centered on participants' personal experience.
  The same topic guide will be used for the first group (epileptic patients) and the second group (relatives group). However, for the third group (bereaved families), the interview guide will be adapted, looking at life experience before death: focusing circumstances, particular events, behaviors or clinical signs which could give alarm.
  Interviews will be digitally recorded

CONTACTS AND LOCATIONS:
Overall Officials: GERALD BOURREL, MD PhD, Study Director — University of Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided